CLINICAL TRIAL: NCT03375502
Title: A Phase II/III, Single-blind(Stage 1), Double-blinded(Stage 2), Randomized, Active-controlled, Dose-escalation(Stage 1), Non-inferiority(Stage 2) Study to Evaluate Immunogenicity and Safety of MG1111 in Healthy Children
Brief Title: A Study of MG1111 in Healthy Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MG1111_P2/3
Record Dates: First submitted 2017-11-28; First posted 2017-12-18 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2017-12

CONDITIONS: Healthy Children
MeSH Terms: interventions — Chickenpox Vaccine; Vaccination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- MG1111(Varicella vaccine) (Experimental): A single injection of 0.5ml MG1111 will be administered subcutaneously at Visit 1
  Interventions: Drug: Varicella Vaccine
- Comparator(Varicella vaccine) (Active Comparator): A single injection of 0.5ml comparator will be administered subcutaneously at Visit 1
  Interventions: Drug: Varicella Vaccine

INTERVENTIONS:
Drug: Varicella Vaccine — The subject will receive investigational product or comparator.
  Other Names: vaccination

SUMMARY:
To assess the safety of MG1111 and to evaluate immunological non-inferiority of MG1111 versus comparator

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 12 months to 12 years.
* Subjects or parent/legal representative willing to provide written informed consent and able to comply with the requirements for the study - Subject able to attend all scheduled visits and to comply with all study procedures
* Negative history of Varicella and varicella vaccine
* Subject in good health, based on medical history and physical examination

Exclusion Criteria:

* Subjects who have a history of Varicella or administration of varicella vaccine
* Subjects who have ahd an acute febrile episode at some time during the 72 hours before administration of investigational product or those who had any symptom suspected to be allergy including systemic rash.

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 814 (Actual)
Dates: Start 2016-11-26 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who achieved seroconversion | 42 days after vaccination

SECONDARY OUTCOMES:
Geometric mean titer(GMT) measured by the FAMA assay | At day 0 and Day 42 post-vaccination
Geometric mean titer(GMT) measured by gpELISA | At day 0 and Day 42 post-vaccination

OTHER OUTCOMES:
Incidence of Local/systemic solicited AEs [Safety] | during the first 7 days after administration of IP
Incidence of Unsolicited AEs [Safety] | Until Day 42 after administration of IP
Incidence of Serious adverse events [Safety] | Until 6 months after administration of IP

CONTACTS AND LOCATIONS:
Locations (1):
- The catholic university of Korea, Seoul st. mary's hospital, Banpo-dong, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No